CLINICAL TRIAL: NCT06053554
Title: Outcome of Two Surgical Methods for IOLImplantation in Eyes With Pseudoexfoliation Syndrome: Lens in the Bag-technique Versus Lens in the Ciliary Sulcus With Optic Capture Technique
Brief Title: Outcome of Two Surgical Methods for IOLImplantation in Eyes With Pseudoexfoliation Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Claudette Abela-Formanek, Univ. Prof., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PEX-2305
Record Dates: First submitted 2023-05-11; First posted 2023-09-25 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Age Related Cataracts; Pseudoexfoliation Syndrome
Keywords: Femtolaser; Sulcus-IOL; Anterior segment; Lens tilt and decentration; Capsular phimoses
MeSH Terms: conditions — Exfoliation Syndrome | interventions — Phacoemulsification

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sulcus (Other): On the day baseline examination, the first eye to be operated is randomised to receive a 3p-IOL implantation in the capsular bag (group 1) or a 3p-IOL haptics in the ciliary sulcus with the IOL optic tucked in the capsular bag (group 2). The second eye to be operated receives the other method. The eye with the lower visual acuity is operated first, in case of identical visual acuity values the for the patient subjective worse eye is operated first. This procedure is clinical standard.
  Interventions: Procedure: Phakoemulsification; Device: Ziemer Z8 Femtolaser; Device: Kowa Avansee Preset
- In the bag (Other): On the day baseline examination, the first eye to be operated is randomised to receive a 3p-IOL implantation in the capsular bag (group 1) or a 3p-IOL haptics in the ciliary sulcus with the IOL optic tucked in the capsular bag (group 2). The second eye to be operated receives the other method. The eye with the lower visual acuity is operated first, in case of identical visual acuity values the for the patient subjective worse eye is operated first. This procedure is clinical standard.
  Interventions: Procedure: Phakoemulsification; Device: Ziemer Z8 Femtolaser; Device: Kowa Avansee Preset

INTERVENTIONS:
Procedure: Phakoemulsification — Femtolaser is used to perform a standard 5.0mm CCC centred on the pupil or limbus and to fragment the lens nucleus toguarantee reproducible results in every eye.After the CCC and nucleus fragmentation the anterior segment is filled with viscoelastics, the rhexis lenticule is removed and hydrodisection of the nucleus is performed. Subsequently phacoemulsification for nucleus and irrigation/aspiration of the lens cortex is performed. The capsular bag and AC is then filled with a cohesive viscoelastic and the IOL is implanted with the haptics in the back or with the haptics in the sulcus. At the end of surgery, the viscoelastic is removed using the irrigation aspiration probe, intracameral antibiotic is instilled, the CCI and paracenteses are hydrated and sealed.
Device: Ziemer Z8 Femtolaser — The femto second laser used for certain steps (capsulorhexis, nucleus fragmentation) of the cataract surgery.
Device: Kowa Avansee Preset — The used 3 piece intra ocular lens

SUMMARY:
The aim of this study is to compare the surgical outcomes of the two IOL implantation methods for eyes with cataract and PEX in a single-center and with highly experienced surgeons. The goal is to acquire relevant information regarding these two IOL implantation techniques, which will help surgeons to decide which approach to choose, ultimately resulting in a benefit for patients with PEX syndrome who require cataract surgery.

The main questions are:

Is there a difference in lens tilt and decentration between the both methods. Is there a difference in the frequency and amount of capsular phimosis between the both methods.

DETAILED DESCRIPTION:
This is a prospective, intraindividual comparative study of two routinely used surgical techniques for IOL implantation in extracapsular cataract surgery. On the day baseline examination, the first eye to be operated is randomised to receive a 3p-IOL implantation in the capsular bag (group 1) or a 3p-IOL haptics in the ciliary sulcus with the IOL optic tucked in the capsular bag (group 2). The second eye to be operated receives the other method. The eye with the lower visual acuity is operated first, in case of identical visual acuity values the for the patient subjective worse eye is operated first. This procedure is clinical standard. Until the point of IOL implantation the surgery is identical in both methods and the surgeon is blinded.

Femtolaser is used to perform a standard 5.0mm CCC centred on the pupil or limbus and to fragment the lens nucleus to guarantee reproducible results in every eye. In case of an insufficient pupil size (smaller than 5.5mm), 2.4mm clear corneal incision and paracenteses are performed prior to laser docking and a pupil expansion device is implanted under anterior segment filling with viscoelastic to enlarge the pupil diameter. After the CCC and nucleus fragmentation the anterior segment is filled with viscoelastics, the rhexis lenticule is removed and hydrodisection of the nucleus is performed. Subsequently phacoemulsification for nucleus and irrigation/aspiration of the lens cortex is performed. The capsular bag and AC is then filled with a cohesive viscoelastic and the IOL is implanted as described above with the haptics in the back or with the haptics in the sulcus. At the end of surgery, the viscoelastic is removed using the irrigation aspiration probe, intracameral antibiotic is instilled, the CCI and paracenteses are hydrated and sealed.

Study investigators are blinded, however the selected method can be visible during the routinely performed slit-lamp examinations. During all evaluation and measuring processes (Evaluation of decentration, tilt, capsular phimoses, surgery time) the investigators are blinded. This study is performed by highly experienced surgeons, who have already performed both methods on a routine basis.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 - 100
* Necessity for bilateral cataract surgery with pseudoexfoliation syndrome
* willing to give informed consent and follow-up the duration of study

Exclusion Criteria:

* Endstage glaucoma
* Christalline lens sub/ luxation
* active inflammatory diseases of the eye

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2030-05 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
The change of lens tilt and decentration from baseline to month 60 postoperatively | Baseline to month 60 postoperatively
  The change of lens tilt and decentration from baseline to month 60 postoperatively, measured by anterior segment optical coherence tomography.
The difference in decentration and tilt between the "in the bag" and the sulcus intra ocular lens implantation method. | Month 60 postoperatively
  The difference in decentration and tilt between the "in the bag" and the sulcus intra ocular lens implantation method at month 60 post operatively, measured by anterior segment optical coherence tomography.

SECONDARY OUTCOMES:
Capsular phimoses | Month 60 postoperatively
  The amount of anterior capsular phimosis and rhexis shrinking, evaluated on anterior segment images.

CONTACTS AND LOCATIONS:
Overall Officials: Claudette ABELA-FORMANEK, Prof. Dr., Principal Investigator — Department for Ophthalmology and Optometry, Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
Publications in peer reviewed journals